CLINICAL TRIAL: NCT06477523
Title: Phase 1b/2 Study of AK104 (Anti-PD1/CTLA4 Bispecific Antibody) in Combination With Etoposide and Carboplatin Plus Low-dose Radiotherapy (LDRT) for the First-line Treatment of Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: Phase 1b/2 Study of LDRT in Combination With AK104 Plus Chemotherapy as First-line Treatment for ES-SCLC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, You Lu, Doctor of Oncology, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-027
Record Dates: First submitted 2024-06-19; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: SCLC, Extensive Stage
MeSH Terms: interventions — Etoposide; Drug Therapy; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDRT+AK104+chemotherapy (Experimental): AK104(IV, D1) + Cisplatin (IV, D1)/Carboplatin (IV, D1) +Etoposide (IV, D1-D3) were administrated on a 21-day cycle for four cycles. Concurrent LDRT (15 Gy/5f) were conducted from D1-D5 in the first cycle. Then pts received LDRT and AK104 maintenance until loss of clinical benefit or unacceptable toxicity.
  Interventions: Drug: AK104; Drug: Etoposide; Drug: Carboplatin; Radiation: low-dose radiotherapy

INTERVENTIONS:
Drug: AK104 — IV infusion
  Other Names: Cadonilimab
Drug: Etoposide — Etoposide intravenous infusion was administered at a dose of 100 mg/m^2 on Days 1, 2, and 3 of each 21-day cycle during the induction phase (Cycles 1-4).
  Other Names: Chemotherapy
Drug: Carboplatin — Carboplatin intravenous infusion to achieve an initial target AUC of 5 mg/mL/min was administered on Day 1 of each 21-day cycle during the induction phase (Cycles 1-4).
  Other Names: Chemotherapy
Radiation: low-dose radiotherapy — The subjects will receive LDRT, from C1D1-C1D5, once a day for 3Gy, until the target dose of 15Gy is achieved (Cycles 1).
  LDRT treatment for primary/mediastinal positive lymph nodes/metastatic lesions during maintenance therapy (C1D1-C1D5, 15Gy).
  Other Names: LDRT

SUMMARY:
Phase Ib/II, open-label, multicentre study to evaluate the efficacy and safety of low-dose radiotherapy (LDRT) combined with AK104 and chemotherapy as first-line treatment for patients with ES-SCLC.

DETAILED DESCRIPTION:
This trial aims to assess the safety and efficacy of a new therapeutic strategy that combines to low-dose radiotherapy combination With AK104 plus etoposide and carboplatin/cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old.
* Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).
* Histologically or cytologically confirmed diagnosis of ES-SCLC per the Veterans Administration Lung Study Group (VALG) staging system.
* No prior treatment for ES-SCLC.
* Measurable disease, as defined by RECIST v1.1.
* Eastern Cooperative Oncology Group performance status ≤ 1.
* Life expectancy ≥ 3 months.
* Adequate hematologic and end-organ function.
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

* Symptomatic or actively progressing Central nervous system metastases.
* Uncontrolled carcinomatous meningitis.
* Uncontrolled severe cancer pain
* Uncontrolled pleural effusion, pericardial effusion or ascites requiring recurrent drainage procedures (once a month or more frequently).
* Uncontrolled or symptomatic hypercalcemia.
* History of autoimmune disease.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (such as bronchiolitis obliterans), drug-induced pneumonia, or idiopathic pneumonia, or evidence of active pneumonia on chest computed tomography (CT) during screening.
* Active Tuberculosis infection.
* Significant cardiovascular disease.
* Major surgical procedure within 28 days prior to enrollment or anticipation of need for major surgical procedure during the course of the study.
* Known additional malignancy that is progressing or requires active treatment.
* Active infection requiring systemic therapy
* Prior allogenic bone marrow transplantation or solid organ transplant.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the participant at high risk for treatment complications.
* Receipt of live attenuated vaccination within 4 weeks prior to the first dose of study treatment, or plan to receive live attenuated vaccine during the study.
* Currently receiving the treatment of hepatitis B virus infection..
* Received approved or under development systematic anti-tumor therapy within 28 days before enrollment
* Previously received immune checkpoint agonists (antibodies to CD137 targets) or immune checkpoint inhibitors (such as anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies, etc.) , immune cell therapy and other treatment of any immune mechanism for tumors
* Treatment with systemic immunosuppressive medications within 1 week prior to enrollment..
* Known allergies or intolerant to test drugs or their excipients; or a known history of severe hypersensitivity reactions to other antibodies.
* Women who are pregnant (positive pregnancy test before medication) or breastfeeding.
* Received chest radiation therapy prior to the first dose.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | 48 months
  The incidence of treatment-related adverse events were measured for determining tolerability and safety. Adverse events (AEs) are evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0). Events of grade 3-5 are defined as moderate and severe adverse events.
Progression free survival at 6 months (PFS-6) | 6 months
  PFS-6 is defined as patient outcomes were evaluated at diagnosis and in the subsets of patients achieving progression-free status at 6 months from diagnosis.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Interval between the date of enrollment and the date of death due to any cause , up to a maximum of approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST V1.1
Progression free survival (PFS) | Interval between the date of enrollment and the date of progressive disease, or death due to any cause (whichever occurs first), up to a maximum of 24 months.
  PFS is defined as the time from the date of first dosing till the first documentation of disease progression (per RECIST v1.1) assessed by the investigator or death due to any cause (whichever occurs first)
PFS Rates at 12 months (PFS-12) | 12 months.
  PFS-6 is defined as patient outcomes were evaluated at diagnosis and in the subsets of patients achieving progression-free status at 12 months from diagnosis.
Overall survival (OS) | Interval between the date of enrollment and the date of progressive disease, or death due to any cause (whichever occurs first), up to a maximum of 24 months.
  OS is defined as the time from randomization to death.
OS Rates at 12 Months (OS-12) | 12 months
  OS-12 is defined as patient outcomes were evaluated at diagnosis and in the subsets of patients survival at 12 months from diagnosis.
OS Rates at 24 Months ( OS-24) | 24 months
  OS-24 is defined as patient outcomes were evaluated at diagnosis and in the subsets of patients survival at 24 months from diagnosis.
Objective Response Rate (ORR) | Interval between the date of enrollment and the date of death from any cause, up to a maximum of 18 months.
  ORR is proportion of subjects with complete response(CR) or partial response(PR). Tumor responses will be evaluated according to RECIST 1.1 criteria. Patients with no tumor assessment after baseline will be classified as non-responders.
Number of participants with adverse events (AEs) | From the subject signs the Informed Consent Form to 90 days after the last dose of study treatment or initiation of other anti-tumor therapy
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product.
  temporally associated with the use of study treatment, whether or not considered related to the study treatment

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - China West Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No